CLINICAL TRIAL: NCT01794169
Title: Azacitidine Compared to Conventional Chemotherapy in Consolidation of Elderly Patients (65 Years or Older) With AML in First Complete Remission
Brief Title: Azacitidine Compared to Conventional Chemotherapy as Consolidation of Elderly Patients With AML
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Karolinska University Hospital (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Stefan Deneberg, M.D, Ph.D., Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWEAML12-a
Record Dates: First submitted 2013-02-13; First posted 2013-02-18 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; Daunorubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azacitidine (Experimental): Azacitidine 75mg/m2/d subcutaneously once daily for 5 days given every 5:th week for 8 cycles.
  Interventions: Drug: Azacitidine
- DA (Active Comparator): Two courses of DA in accordance with the Swedish National treatment program (reduced doses):
  In case one induction course was given:
  First consolidation course: daunorubicin 45 mg/m2 x 1 (iv infusion) day 1-3 and cytarabine 1000 mg/m2 x 2 (iv infusion) day 1-4.
  Second consolidation course: daunorubicin 45 mg/m2 x 1( iv infusion) day 1-2 and cytarabine 200 mg x 2 (fixed dose sc injection) day 1- 5.
  In case two induction courses were given:
  First consolidation course: daunorubicin 45 mg/m2 x 1( iv infusion) day 1-2 and cytarabine 200 mg x 2 (fixed dose sc injection) day 1- 5.
  Second consolidation course: cytarabine 200mg x 2 (fixed dose sc injection) day 1-5.
  Interventions: Drug: DA

INTERVENTIONS:
Drug: Azacitidine
  Other Names: Vidaza
  Arms: Azacitidine
Drug: DA
  Other Names: Daunorubicin; Cytarabine; Ara-C
  Arms: DA

SUMMARY:
The purpose of this study is to determine whether Azacitidine consolidation is superior to standard DA consolidation treatment of acute myeloid leukemia in first complete remission in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects >65 years of age at the time of signing the informed consent form
2. A confirmed diagnosis of AML according to the 2008 WHO classification

   * This includes: Bone marrow aspirate with a good clot or biopsy for morphology, flow cytometry, cytogenetic analysis, and in case of normal cytogenetics, molecular genetic analyses including FLT3-ITD, NPM-1 and CEBP A
   * Bio-banking of leukemic cells at diagnosis performed (according to guidelines of the Swedish National AML biobank).
3. A documented CR or CRp achieved after one or two induction courses.

Exclusion Criteria:

1. Subjects who are not considered to be candidates to complete the consolidation therapy due to medical or psychological reasons.
2. Subjects who have taken any investigational drugs or participated in an interventional clinical trial within 30 days prior to screening.
3. Patients with acute promyelocytic leukemia
4. Patients with t(8;21) or inv(16)
5. CNS leukemia
6. Patients with a previous diagnosis of MDS, i.e. AML preceded by a diagnosed MDS
7. Subjects who are candidates for allogeneic stem cell transplantation (SCT)
8. Another cancer diagnosis with a life expectancy of less than two years

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-09 (Actual); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Leukemia free survival | One year

SECONDARY OUTCOMES:
Overall survival | Two years
Treatment related morbidity and mortality | Two years
Severe Adverse Events (SAE) | Two months after the last course of consolidation
  SAE as defined by CTCAE
Number of days admitted in hospital | 12 months from start of consolidation treatment
Quality of life | Until 24 months from start of consolidation treatment
  EORTC QLQ C30
Number of participants with AE grade 3 or more | Until two months after the last course of consolidation
  AE:s graded according to CTCAE
Number of consolidation courses actually given within the study | One year

OTHER OUTCOMES:
Molecular analyses | Two years
  Analysis of a broad spectrum of molecular and cellular events relating to the epigenetic status of the malignant cells. These events will be used to identify biomarkers for successful consolidation and to address whether AML cases that relapse while on the study are molecularly and epigenetically different between those given azacitidine or DA consolidation
Leukemia free survival (LFS) | One year
  Analysis whether cytogenetic and molecular aberrations at diagnosis will predict for better LFS with either Azacitidine or standard DA consolidation.

CONTACTS AND LOCATIONS:
Overall Officials: Per Bernell, M.D., Ph.D., Principal Investigator — Karolinska University Hospital; Stefan Deneberg, M.D., Ph.D., Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Solna, Stockholm, Sweden